CLINICAL TRIAL: NCT00299767
Title: Phase I Study of Sequential Cord Blood Transplants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Karen Ballen, Director, Leukemia Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-061
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Lymphoma; Leukemia; Multiple Myeloma; Myelodysplastic Syndrome
MeSH Terms: conditions — Lymphoma; Leukemia; Multiple Myeloma; Myelodysplastic Syndromes

INTERVENTIONS:
Procedure: sequential cord blood transplantation — Infused on Day 0

SUMMARY:
The purpose of this study is to determine the safety of sequential cord blood transplantation (2 cord blood units) for patients who have diseases that are capable of being cured by allogeneic stem cell transplant but do not have a matched family or volunteer unrelated donor.

DETAILED DESCRIPTION:
Eligible patients will receive conditioning therapy with fludarabine 30 mg/m2/day x 6 days, melphalan 100 mg/m2/day x 1 day, rabbit antithymocyte globulin 1.5 mg/kg/day x 4 days. GVHD prophylaxis will consist of cyclosporine starting on day -1 and mycophenolate mofetil starting on day 0. Sequential cord blood units will be infused on Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Disease Status: NHL, HD, or MM refractory to chemotherapy or relapsed; CLL Rai Stage III/IV, or lymphocyte doubling time of 6 months, or Stage I/II resistant to 2 chemotherapy regimens; AML or ALL in second or subsequent remission or in first remission with adverse cytogenetics or antecedent hematologic disorder
* Estimated disease-free survival of less than one year
* ECOG performance status of 0, 1, 2
* Lack of 6/6 or 5/6 HLA matched related or 6/6 matched unrelated donor, or a donor is not available within the time frame necessary to perform a potentially curative stem cell transplant
* 4/6 or greater HLA A, B, CRB1 cord blood units with a combined nucleated cell dose from of > 3.7 x 10(7) NC/kg

Exclusion Criteria:

* Cardiac disease: symptomatic congestive hearth failure or RVG or echocardiogram determined left ventricular ejection fraction of < 45%, active angina pectoris, or uncontrolled hypertension
* Pulmonary Disease: severe chronic obstructive lung disease, or symptomatic restrictive lung disease, or corrected DLCO of < 50%
* Renal disease: serum creatinine > 2.0 mg/dl
* Hepatic disease: serum bilirubin > 2.0 mg/dl (except in the case of Gilbert's syndrome), SGPT or SGOT > 3 x normal
* Neurologic disease: symptomatic leukoencephalopathy, active DNS malignancy or other neuropsychiatric abnormalities believed to preclude transplantation
* HIV antibody or Hepatitis B surface antigen positivity
* Uncontrolled infection
* Pregnancy or breast-feeding mother

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-05; Primary Completion 2005-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the 100-day transplant-related (non-relapse) mortality, including relapse-related mortality associated with Grade 4 toxicity. | 3 years

SECONDARY OUTCOMES:
To evaluate the 6 month transplant related (non-relapse) mortality. | 3 years
To evaluate the days to neutrophil engraftment (ANC > 500). | 3 years
To evaluate the days of platelet engraftment (platelet count > 20K unsupported). | 3 years
To evaluate the risk of acute and chronic graft versus host disease. | 3 years
To evaluate percent donor chimerism - contribution of each cord unit. | 3 years
To evaluate relapse rate.
To evaluate overall survival.
To evaluate transfusion support needed to cord blood transplant recipients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ballen, M.D., Principal Investigator — Massachusetts General Hospital, Harvard University; Joseph Antin, M.D., Principal Investigator — Dana Farber Cancer Institute, Harvard Univeristy; David Avigan, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts